CLINICAL TRIAL: NCT00663260
Title: A Multicenter, Double-Blind, Placebo-Controlled, Parallel Group, Randomized, Phase 2/3 Trial to Evaluate the Glycemic Efficacy, Renal Safety, Pharmacokinetics, and Pharmacodynamics of Dapagliflozin in Subjects With Type 2 Diabetes Mellitus and Moderate Renal Impairment Who Have Inadequate Glycemic Control
Brief Title: Glycemic Efficacy and Renal Safety Study of Dapagliflozin in Subjects With Type 2 Diabetes Mellitus and Moderate Renal Impairment
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MB102-029
Record Dates: First submitted 2008-04-18; First posted 2008-04-22 (Estimated); Results first posted 2017-02-10 (Actual); Last update posted 2017-02-10 (Actual); Status verified 2016-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dapagliflozin (10 mg) (Active Comparator)
  Interventions: Drug: Dapagliflozin
- Dapagliflozin (5 mg) (Active Comparator)
  Interventions: Drug: Dapagliflozin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — Tablets, Oral, 10 mg, Once Daily, 104 weeks
  Other Names: BMS-512148
  Arms: Dapagliflozin (10 mg)
Drug: Dapagliflozin — Tablets, Oral, 5 mg, Once Daily, 104 weeks
  Other Names: BMS-512148
  Arms: Dapagliflozin (5 mg)
Drug: Placebo — Tablets, Oral, 0 mg, Once Daily, 104 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether dapagliflozin is effective in the treatment of type 2 diabetes in subjects with poor blood sugar control and moderate renal impairment

DETAILED DESCRIPTION:
All eligible subjects will receive a single-blind placebo medication during a 1-week lead-in period prior to randomization. All arms may include the addition of open label medication described (as needed for rescue based on protocol specific criteria). Rescue medication is defined as the addition of an approved, appropriate antihyperglycemic agent, except metformin, used according to conventional standards of care, to treat hyperglycemia, which may therefore allow the subject to remain in the trial

ELIGIBILITY:
Inclusion Criteria:

* Males and females, ≥18 years old, with type 2 diabetes and with inadequate glycemic control
* Clinical diagnosis of moderate renal impairment

Exclusion Criteria:

* AST and /or ALT > 3.0 times the upper limit of normal
* Serum total bilirubin > 1.5 times ULN
* Symptoms of severely uncontrolled diabetes
* Currently unstable or serious cardiovascular, hepatic, hematological, oncological, endocrine, psychiatric, or rheumatic diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 631 (Actual)
Dates: Start 2008-06; Primary Completion 2009-12 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (87):
- United States (34):
  - Vista Medical Research, Inc., Mesa, Arizona
  - Valley Research, Fresno, California
  - Marin Endocrine Care & Research, Inc., Greenbrae, California
  - Office Of Richard Cherlin, Md, Los Gatos, California
  - Diabetes Medical Center Of California, Northridge, California
  - Apex Research Of Riverside, Riverside, California
  - La Biomed At Harbor Ucla Med Ctr., Torrance, California
  - Endocrine Associates Of The Rockies, Denver, Colorado
  - Panhandle Family Care Associates, Marianna, Florida
  - Genesis Clinical Research, Tampa, Florida
  - Endocrine Research Solutions, Inc., Roswell, Georgia
  - Twin Cities Clinical Research, Brooklyn Center, Minnesota
  - Kcva Medical Center Research Svc (151), Kansas City, Missouri
  - Va Nebraska-Western Iowa Health Care System (Nwihcs), Omaha, Nebraska
  - University Of Medicine And Dentistry Of New Jersey, Voorhees Township, New Jersey
  - Winthrop University Hospital, Mineola, New York
  - Slocum-Dickson Medical Group, Pllc, New Hartford, New York
  - Community Health Care Of Manchester, Akron, Ohio
  - Center For Thyroid Diseases And Endocrinology, Beachwood, Ohio
  - Physician Research, Inc., Zanesville, Ohio
  - Univ Of Oklahoma Health Science Center, Oklahoma City, Oklahoma
  - Rogue Valley Clinical Research, Medford, Oregon
  - Drexel University College Of Medicine, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Low Country Internal Medicine Of Sc, Pa, Charleston, South Carolina
  - Carolina Health Specialists, Myrtle Beach, South Carolina
  - Palmetto Clinical Research, Summerville, South Carolina
  - Research Institute Of Dallas, Dallas, Texas
  - Westbury Medical Clinic P.A., Houston, Texas
  - The Strelitz Diabetes Center, Norfolk, Virginia
  - Capital Clinical Research Center, Olympia, Washington
  - Cedar Research Llc, Tacoma, Washington
  - Aurora Advanced Healthcare, Milwaukee, Wisconsin
  - Zablocki Veterans Affairs Medical Center, Milwaukee, Wisconsin
- Argentina (6):
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, Capital Federal, Buenos Aires
  - Local Institution, Mar del Plata, Buenos Aires
  - Local Institution, Zárate, Buenos Aires
  - Local Institution, Córdoba, Córdoba Province
  - Local Institution, Salta, Salta Province
- Australia (4):
  - Local Institution, Camperdown, New South Wales
  - Local Institution, St Leonards, New South Wales
  - Local Institution, Woollongong, New South Wales
  - Local Institution, Launceston, Tasmania
- Canada (9):
  - Local Institution, Calgary, Alberta
  - Local Institution, Winnipeg, Manitoba
  - Local Institution, Barrie, Ontario
  - Local Institution, Thornhill, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Gatineau, Quebec
  - Local Institution, Laval, Quebec
  - Local Institution, Sherbrooke, Quebec
  - Local Institution, Regina, Saskatchewan
- Denmark (3):
  - Local Institution, Copenhagen Nv
  - Local Institution, Gentofte Municipality
  - Local Institution, Hvidovre
- France (4):
  - Local Institution, Besançon
  - Local Institution, Brest
  - Local Institution, Paris
  - Local Institution, Poitiers
- India (5):
  - Local Institution, Indore, Madhya Pradesh
  - Local Institution, Pune, Maharashtra
  - Local Institution, Bangalore
  - Local Institution, Chennai
  - Local Institution, Rajasthan
- Italy (8):
  - Local Institution, Chieri
  - Local Institution, Chieti Scalo
  - Local Institution, Modena
  - Local Institution, Padua
  - Local Institution, Perugia
  - Local Institution, Pisa
  - Local Institution, Roma
  - Local Institution, Siena
- Mexico (5):
  - Local Institution, Durango, Durango
  - Local Institution, Celaya, Guanajuato
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Df, Mexico City
  - Local Institution, Monterrey, Nuevo León
- Peru (3):
  - Local Institution, Arequipa, Arequipa
  - Local Institution, Lima, Lima Province
  - Local Institution, Lima Cercado, Lima region
- Puerto Rico (2):
  - Local Institution, Caguas
  - Local Institution, San Juan
- Local Institution, Singapore, Singapore
- Spain (3):
  - Local Institution, Barcelona
  - Local Institution, San Sebastian de Los
  - Local Institution, Vizcaya

REFERENCES:
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818
- [Derived] Fioretto P, Stefansson BV, Johnsson E, Cain VA, Sjostrom CD. Dapagliflozin reduces albuminuria over 2 years in patients with type 2 diabetes mellitus and renal impairment. Diabetologia. 2016 Sep;59(9):2036-9. doi: 10.1007/s00125-016-4017-1. Epub 2016 Jun 15. No abstract available. PMID 27306615
- [Derived] Kohan DE, Fioretto P, Tang W, List JF. Long-term study of patients with type 2 diabetes and moderate renal impairment shows that dapagliflozin reduces weight and blood pressure but does not improve glycemic control. Kidney Int. 2014 Apr;85(4):962-71. doi: 10.1038/ki.2013.356. Epub 2013 Sep 25. PMID 24067431
- See also: Publication — http://rd.springer.com/article/10.1007%2Fs00125-016-4017-1
- See also: Publication long-term — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3973038/
- See also: MB102029_Redacted_CSR_synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3639&filename=MB102029_Redacted_CSR_synopsis.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 631 participants enrolled, 276 completed a qualification period. Of these 276 participants, 252 were randomized and received treatment. Of these 252 participants, 204 completed double-blind treatment period.
Groups:
- Placebo: Participants received dapagliflozin matching placebo once daily for up to 24 weeks (Subjects were to continue their original pre-enrollment anti-diabetic therapy; may include the addition of open-label anti-diabetic therapy as rescue)
- Dapagliflozin 5 mg: Participants received dapagliflozin 5 mg once daily for up to 24 weeks (Subjects were to continue their original pre-enrollment anti-diabetic therapy; may include the addition of open-label metformin as rescue)
- Dapagliflozin 10 mg: Participants received dapagliflozin 10 mg once daily for up to 24 weeks (Subjects were to continue their original pre-enrollment anti-diabetic therapy; may include the addition of open-label metformin as rescue)
Period: Overall Study
Arm/Group | Placebo | Dapagliflozin 5 mg | Dapagliflozin 10 mg
Started | 84 | 83 | 85
Completed | 63 | 72 | 69
Not Completed | 21 | 11 | 16
Not completed — Lack of Efficacy | 2 | 0 | 0
Not completed — Adverse Event | 12 | 7 | 6
Not completed — Withdrawal by Subject | 3 | 1 | 6
Not completed — Death | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — non-compliance, not met criteria, etc. | 3 | 2 | 3

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study medication
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dapagliflozin 5 mg | Dapagliflozin 10 mg | Total
Number analyzed (Participants) | 84 | 83 | 85 | 252
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67 (8.6) | 66 (8.9) | 68 (7.7) | 67 (8.4)
Age, Customized [Number; unit: Participants]
  Younger than 65 years | 36 | 39 | 29 | 104
  65 years and older | 48 | 44 | 56 | 148
Sex/Gender, Customized [Number; unit: Participants]
  Male | 53 | 55 | 56 | 164
  Female | 31 | 28 | 29 | 88
Race/Ethnicity, Customized [Number; unit: Participants]
  WHITE | 69 | 65 | 77 | 211
  BLACK OR AFRICAN AMERICAN | 1 | 7 | 4 | 12
  ASIAN | 6 | 4 | 3 | 13
  OTHER | 8 | 7 | 1 | 16
Weight [Mean (Standard Deviation); unit: kg] | 89.61 (20.046) | 95.23 (20.909) | 93.25 (17.309) | 92.69 (19.529)
Pre-Enrollment Anti-Hyperglycemic Therapy [Number; unit: Participants]
  INSULIN-BASED REGIMEN | 55 | 54 | 55 | 164
  SULFONYLUREA-BASED REGIMEN | 21 | 21 | 21 | 63
  THIAZOLIINEDIONE-BASED REGIMEN | 1 | 1 | 2 | 4
  OTHER REGIMEN | 7 | 7 | 7 | 21

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change From Baseline in Hemoglobin A1C (HbA1c) at Week 24 (Last Observation Carried Forward [LOCF]
Description: HbA1c was measured as percent of hemoglobin by a central laboratory. Data after rescue medication was excluded from this analysis. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. HbA1c measurements were obtained during the qualification and lead-in periods and on Day 1 and Weeks 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, and 24 in the double-blind period.
Time Frame: From Baseline to Week 24
Population: All randomized participants who received study medication and had nonmissing HbA1c values at baseline and Week 24 (LOCF)
Measure: Mean (Standard Error); unit: % of hemoglobin
Arm/Group | Placebo | Dapagliflozin 5 mg | Dapagliflozin 10 mg
Number analyzed (Participants) | 82 | 83 | 82
% of hemoglobin | -0.32 (0.1701) | -0.41 (0.1701) | -0.44 (0.1708)
Statistical Analysis 1: Comparison: Placebo vs Dapagliflozin 5 mg; Test type: Superiority or Other; p = 0.561, ANCOVA — Primary endpoints were tested at alpha=0.027 applying Dunnett's adjustment; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.37 to 0.20], Standard Error of Mean 0.1448
Statistical Analysis 2: Comparison: Placebo vs Dapagliflozin 10 mg; Test type: Superiority or Other; p = 0.435, ANCOVA — Primary endpoints were tested at alpha=0.027 applying Dunnett's adjustment; Mean Difference (Final Values) = -0.11, 95% CI 2-sided [-0.40 to 0.17], Standard Error of Mean 0.1457

2. Secondary Outcome: Adjusted Mean Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24 (Last Observation Carried Forward [LOCF])
Description: Secondary endpoints were tested using sequential testing procedure and are presented in hierarchical order. Fasting plasma glucose was measured as milligrams per deciliter(mg/dL) by a central laboratory. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. FPG measurements were obtained during the qualification and lead-in periods and on Day 1 and Weeks 1, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, and 24 in the double-blind period
Time Frame: From Baseline to Week 24
Population: All randomized participants who received study medication and had nonmissing FPG values at baseline and Week 24 (LOCF)
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Dapagliflozin 5 mg | Dapagliflozin 10 mg
Number analyzed (Participants) | 83 | 83 | 85
mg/dL | 8.4 (9.621) | -5.2 (9.548) | -0.6 (9.524)
Statistical Analysis 1: Comparison: Placebo vs Dapagliflozin 5 mg; Test type: Superiority or Other; ANCOVA — Secondary endpoints were tested following a sequential testing procedure at alpha=0.05; secondary efficacy analyses were not tested since the primary endpoint was not significant; Mean Difference (Final Values) = -13.6, 95% CI 2-sided [-29.7 to 2.4], Standard Error of Mean 8.142
Statistical Analysis 2: Comparison: Placebo vs Dapagliflozin 10 mg; Test type: Superiority or Other; ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -9.0, 95% CI 2-sided [-25.0 to 7.0], Standard Error of Mean 8.136

3. Secondary Outcome: Adjusted Mean Change From Baseline in Total Body Weight (kg) at Week 24 (Last Observation Carried Forward [LOCF])
Description: Secondary endpoints were tested using sequential testing procedure and are presented in hierarchical order. Adjusted mean change from baseline in total body weight at Week 24 (or the last postbaseline measurement prior to Week 24 if no Week 24 assessment was available was determined. Data after rescue medication was excluded from this analysis. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. Body weight measurements were obtained during the qualification and lead-in periods and on Day 1 and Weeks 1, 2, 4, 8, 12, 16, 20, and 24 of the double-blind period.
Time Frame: From Baseline to Week 24
Population: All randomized participants who received study medication and had nonmissing body weight values at baseline and Week 24 (LOCF)
Measure: Mean (Standard Error); unit: kg
Arm/Group | Placebo | Dapagliflozin 5 mg | Dapagliflozin 10 mg
Number analyzed (Participants) | 84 | 83 | 85
kg | 0.27 (0.4872) | -1.54 (0.4815) | -1.89 (0.4693)
Statistical Analysis 1: Comparison: Placebo vs Dapagliflozin 5 mg; Test type: Superiority or Other; ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -1.81, 95% CI 2-sided [-2.68 to -0.94], Standard Error of Mean 0.4435
Statistical Analysis 2: Comparison: Placebo vs Dapagliflozin 10 mg; Test type: Superiority or Other; ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -2.16, 95% CI 2-sided [-3.03 to -1.29], Standard Error of Mean 0.4395

ADVERSE EVENTS:
Time Frame: Onset on or after the first date of double-blind treatment and on or prior to the last day of double-blind treatment 24 weeks plus 4 days for non-serious adverse event; plus 30 days for serious adverse event.
Arm/Group | Placebo | Dapagliflozin 5 mg | Dapagliflozin 10 mg
Serious Adverse Events (participants affected / at risk) | 9/84 | 7/83 | 12/85
Other Adverse Events (participants affected / at risk) | 39/84 | 45/83 | 42/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=84) | Dapagliflozin 5 mg (N=83) | Dapagliflozin 10 mg (N=85)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
CEREBRAL INFARCTION (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
RETINAL DETACHMENT (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
CELLULITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
HEART RATE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
HYPOTENSION (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
INGUINAL HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
CHEST PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0)
OEDEMA (General disorders) | 1 (1) | 0 (0) | 0 (0)
HYPERSENSITIVITY (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
TRAUMATIC BRAIN INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
SPONDYLOLISTHESIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
TENDON DISORDER (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
BALANOPOSTHITIS (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=84) | Dapagliflozin 5 mg (N=83) | Dapagliflozin 10 mg (N=85)
POLLAKIURIA (Renal and urinary disorders) | 3 (3) | 5 (7) | 10 (12)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 8 (9) | 8 (10)
DIARRHOEA (Gastrointestinal disorders) | 3 (3) | 3 (4) | 8 (9)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 3 (5) | 3 (3) | 7 (8)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 3 (5) | 7 (7)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 (4) | 3 (4) | 6 (7)
DIZZINESS (Nervous system disorders) | 4 (4) | 10 (14) | 5 (5)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 10 (16) | 7 (9) | 5 (6)
HYPERTENSION (Vascular disorders) | 5 (6) | 1 (1) | 5 (5)
NASOPHARYNGITIS (Infections and infestations) | 5 (8) | 6 (6) | 4 (5)
OEDEMA PERIPHERAL (General disorders) | 4 (4) | 8 (10) | 4 (6)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 5 (6) | 5 (5) | 2 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 6 (7) | 7 (8) | 2 (2)
MICTURITION URGENCY (Renal and urinary disorders) | 0 (0) | 5 (5) | 2 (3)
GASTROENTERITIS (Infections and infestations) | 5 (6) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No